CLINICAL TRIAL: NCT05973162
Title: Effects of Virtual Reality as an Adjunctive to Transverse Friction Massage in Pediatric Burn Patients
Brief Title: Effects of Virtual Reality in Pediatric Burn Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01651 Lareb Sattar
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Burns Elbows; Pediatric ALL
Keywords: Virtual Reality; Pediatric burn patients,; transverse friction massage; Elbow burn injuries
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Virtual Reality training (Active Comparator): Virtual Reality + Conventional PT
  Interventions: Other: Virtual Realty Training
- Transverse friction massage (TFM) (Experimental): Transverse friction massage (TFM)+ Conventional PT
  Interventions: Other: Transverse friction massage (TFM)

INTERVENTIONS:
Other: Virtual Realty Training — They would be receiving treatment as follow:
  Virtual Reality is a technology that aims to completely immerse the user inside the computer generated world, giving the impression to the user that they have "stepped inside" the synthetic world. RA mobile phone , head mounted display (HMD) will be used and videos of patient's interest will be played on phone which will create a 3D world around the patient.
  And while watching conventional physical therapy will be performed side by side.
  Conventional PT including range of motion exercises of elbow region including flexion, extension, supination, pronation, stretching and strengthening exercises of elbow muscles. Frequency: 10 reps with 5 sec hold for 3 times/week for 2 weeks Intensity: moderate-high intensity (depending on pain tolerance) Time: 10 mins Type: Strengthening Exercises
  Arms: Virtual Reality training
Other: Transverse friction massage (TFM) — They would be receiving treatment as follow:
  Transverse friction massage (Soft tissue mobilization technique) on the surrounding burn region for 5-10min in intervals. Frequency: 3 times/week for 2 consecutive weeks. Intensity: moderate intensity (pain free) Time: 10 mins Conventional PT including range of motion exercises of elbow region including flexion, extension, supination, pronation, stretching and strengthening exercises of elbow muscles. Frequency: 10 reps with 5 sec hold for 3 times/week for 2 weeks Intensity: moderate-high intensity (depending on pain tolerance) Time: 10 mins Type: Strengthening Exercises
  Arms: Transverse friction massage (TFM)

SUMMARY:
The aim of this randomized controlled trial is to find the effectiveness of Virtual reality as an adjunctive to transverse friction massage in pediatric burn patients for reducing pain, anxiety and enhancing elbow range of motion.

DETAILED DESCRIPTION:
A burn injury is damage to the skin or other body parts caused by heat, chemicals, electricity, radiation, or friction.Pain or discomfort, redness and swelling, blistering, peeling skin, scarring , difficulty breathing, shock in cases of severe burn, fever as a complication of burn, anxiety and depression are some main signs and symptoms after burn injuries. Upper limb burn injuries are more common as compared to lower limb , trunk or head and neck. Physical therapy plays an important role in reducing pain and improving range of motion and prevention of contractures formation after burn injuries.

Virtual Reality training (VR) uses a computer-generated simulation of a three-dimensional environment that can be interacted with in a seemingly real or physical way. In the context of burn injuries, VR can be used as a distraction technique during wound care procedures or as an adjunct to pain management, and reduction of anxiety level.

Transverse friction massage Therapy is a Cyriax technique , is applied by the fingers directly to the lesion and transverse to the direction of fibers.Pressure is applied with the ball of the practitioners thumb or fingers to the patient's skin or muscles. Friction massage applied correctly will quickly result in analgesic effect over the treated area. Friction prevents the adhesion formations as a result leads to improvement of range of motion , prevention of contractures formation as well as pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Willingly participated in the study.
* Age group:6-18.
* Gender: both Male and Female
* Acute burn injuries of elbow region (grade 2)
* Superficial wounds healing phase( 5-10) days
* TBSA is less than 20%

Exclusion Criteria

* Motion sickness
* History of seizure activity
* Burns on body region that impede use of VR equipment (ears, eyes, head)
* Deep burn (Grade 3,4)
* Fractures

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-03-28 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Mayo Elbow Performance Index | 2 weeks
  MEPI is an instrument used to test the limitations, caused by pathology, of the elbow during activities of daily living (ADL). This specific test uses 4 subscales:
  * Pain,
  * Range of Motion
  * Stability
  * Daily Function The clinical information is rated based on a 100 points scale.
  * <60 - poor
  * 60-74 - fair
  * 75-89 - good
  * 90-100 - excellent

SECONDARY OUTCOMES:
Burn Specific Pain Anxiety Scale (BSPAS) | 2 weeks
  The BSPAS is a 9 item self report scale for the assessment of pain related and anticipatory anxiety in burn patients. The items are scored on a 100 mm visual analog line with two reference points given values of 0 and 100. The reference points are identified by these numbers, and also by the expressions 'not at all' and 'the worst imaginable way'. There is no middle ranged reference position or 'neutral' point on this visual analog line.
Goniometer | 2 weeks
  It is an instrument that measures the available range of motion at a joint.

CONTACTS AND LOCATIONS:
Overall Officials: Kinza Anwar, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Burn units of Rawalpindi/Islamabad (PIMS hospital, Max Health hospital), Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No